CLINICAL TRIAL: NCT05493358
Title: Long-term Outcomes of Open Versus Laparoscopic Distal Gastrectomy for T4a Gastric Cancer: a Propensity Score-matched Cohort Study
Brief Title: Long-term Outcomes of Open Versus Laparoscopic Distal Gastrectomy for T4a Gastric Cancer
Status: Completed | Type: Observational
Sponsor: University Medical Center Ho Chi Minh City (UMC) (Other)
Responsible Party: Sponsor
Other Study IDs: 71/GCN-HĐĐĐ
Record Dates: First submitted 2022-08-04; First posted 2022-08-09 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2022-08

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Open distal gastrectomy: An incision of 15~20 cm length is made in the abdominal midline . Standard distal gastrectomy and omentectomy will be performed with D2 lymph node dissection (around common hepatic artery, celiac artery, proximal part of splenic artery, proper hepatic artery) . As a general rule, Billroth I, Billroth II or Roux en Y method was used for gastric reconstruction.
- Laparoscopic distal gastrectomy: 5 trocar were used. The gastrocolic ligament was divided along the border of the transverse colon. ligating the left gastroepiploic vessels to remove group 4sb.
  The right gastroepiploic vein was divided and the right gastroepiploic and the inferior pyloric artery were vascularized and cut at their origin from the gastroduodenal artery, just above the pancreatic head, to dissect group 6.
  The dissection was continued along the hepatoduodenal ligament to removed group 5 and group 12a and along the common hepatic artery to remove group 8a and along the celiac axis to remove group 9.
  The left gastric vein was prepared and separately divided and then the left gastric artery was vascularized to remove group 7.
  The dissection was continued upward along the proximal branches of splenic vessels to remove group 11p and along the lesser curvature to remove group 1,3.
  As a general rule, Billroth I, Billroth II or Roux en Y method was used for gastric reconstruction.
  Interventions: Procedure: Laparoscopic distal gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic distal gastrectomy — Distal gastrectomy and standard D2 lymphadenectomy
  Groups: Laparoscopic distal gastrectomy

SUMMARY:
There are more than 75% of patients with gastric cancer who are diagnosed in advanced stage in Vietnam, most of cases in T4a. The purpose of this study was to compare short- and long- term outcomes of open and laparoscopic distal gastrectomy for gastric adenocarcinoma in surgical T4A stage.

DETAILED DESCRIPTION:
Gastric cancer is one of the most common cancers in Vietnam . Despite recent advances in multimodality treatment and targeted therapy, surgery remains the first option of treament for this disease. For resectable gastric cancer, complete removal of macroscopic and microscopic lesions and/or combined resections and also regional or extended lymphadenectomy should represent worldwide now.

Laparoscopic gastrectomy for locally advanced gastric cancer AGC have commonly used for treatment of AGC, especially in Japan, Korea and China. However, the real role of laparoscop for treament of (AGC) is still controversial in term of technical feasibility, safety and oncologic aspect for T4a stage.

Paragastric inflammatory strands may occur in T4a tumor so that laparoscopic technique is difficult to radically perform. Peritoneal seeding of malignant cells, intra- and postoperative complications, trocarts metastasis may risk during procedures. Despite, some studies have demonstrated the safety and the short-term benefits of LG for T4a gastric cancer, the number of these studies and sample sizes have been still inadequate to give good evidence for applying it. and long-term oncologic outcomes There are more than 75% of patients with gastric cancer who are diagnosed in advanced stage in Vietnam, most of cases in T4a. The purpose of this study was to compare short- and long- term outcomes of open and laparoscopic distal gastrectomy for gastric adenocarcinoma in surgical T4A stage.

ELIGIBILITY:
Inclusion Criteria:

* patients with histologically confirmed adenocarcinoma of the stomach, surgical staging of sT4aN0-3M0 according to the 7th edition of the American Joint Committee on Cancer/Union Internationale Contre le Cancer (AJCC/UICC) staging system

Exclusion Criteria:

* intraoperatively detected bulky lymph nodes
* inadequate lymphadenectomy (D0, D1, D1+)
* macroscopic residual tumor (R2)
* an American Society of Anaesthesiology (ASA) score of > IV
* concurrent cancer or history of previous other cancers
* previous gastrectomy
* neoadjuvant chemotherapy
* complications such as bleeding or perforation required emergency gastrectomy.

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients with surgical T4a (sT4a) gastric adenocarcinoma at the lower or middle third of the stomach who underwent ODG or LDG plus lymphadenectomy between January 2013 and December 2020 at the Gastro-intestinal Surgical Department of the University Medical Center at Ho Chi Minh City, Vietnam
Sampling Method: Non-Probability Sample
Enrollment: 472 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
5 year overall survival by Kaplan Mayer | 5 year after surgery
  The percentage of people in this study who are alive five years after surgery.
5 year disease-free survival by Kaplan Mayer | 5 year after surgery
  The percentage of people in this study who are alive without recurrence/metastasis five years after surgery.

SECONDARY OUTCOMES:
1 year overall survival by Kaplan Mayer | 1 year after surgery
  The percentage of people in this study who are alive one years after surgery.
3 year overall survival by Kaplan Mayer | 3 year after surgery
  The percentage of people in this study who are alive one years after surgery.
1 year disease-free survival by Kaplan Mayer | 1 year after surgery
  The percentage of people in this study who are alive without recurrence/metastasis one years after surgery.
3 year disease-free survival by Kaplan Mayer | 3 year after surgery
  The percentage of people in this study who are alive without recurrence/metastasis one years after surgery.
operative morbidity | 30 days after surgery
  The overall rate of postoperative complications
operative time | intraoperative
  The duration of a surgical procedure in minutes.
operative blood loss | intraoperative
  The amount of blood lost during procedure
time to flatus | 30 days after surgery or until mortality ]
  Number of days from date of surgery until date of flatus
Postoperative hospital length of stay | 30 days after surgery or until mortality
  Number of days from date of surgery until date of discharge or mortality
The percentage of complications with Clavien-Dindo | 30 days after surgery
  The percentage of complication grade by Clavien-Dindo classification
The percentage of pattern of recurrence/metastasis | 5 year after surgery
  The percentage of pattern of recurrence/metastasis during follow up period

CONTACTS AND LOCATIONS:
Overall Officials: Long D. Vo, MD PhD., Principal Investigator — University Medical Center HCMC, Vietnam
Locations (1):
- University Medical Center Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No